CLINICAL TRIAL: NCT02295579
Title: Vaginal Colonization After Treatment With Lactobacillus in Women With BV or Candida Will That Increase the Cure Rate After Treatment With Clindamycin for BV and Flucnazole for Candida
Brief Title: Will Lactobacillus Increase Cure Rate After Treatment of Bacterial Vaginosis and Chronic Vulvovaginal Candida
Status: Completed | Type: Observational
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Per-Goran Larsson, Professor Consultat, Skaraborg Hospital
Other Study IDs: 24580-53750
Record Dates: First submitted 2014-10-30; First posted 2014-11-20 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Lacteol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: lactobacillus (EcoVag) — Probiotic human lactobacillus (L. gasseri and L rahmnosus)

SUMMARY:
From the earlier studies the investigators have treated women with bacterial vaginosis and cronic vulvovaginal candida. The investigators have then treated them with laktobacilli 10 days for 2 month. The investigators will continue to follow them and investigate if treatment with lactobacilli every week for 6 month will increase cure rate.

DETAILED DESCRIPTION:
Clinical diagnosis of bacterial vaginosis using air dried smears combined with Hay/Ison classification. Test of cure every month or every menstrual cycle using self taken smears. The cure will be if the woman are in group 1 according to Hay/Ison classification. This will also allow us to use molecular diagnosis of BV to test cure and compare this with hay/Ison.

Test of cure for candida patiens are no visibel candida on wet smear and free of symtoms of candida.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bacterial vaginosis according to Hay/Ison or with candida diagnosed with wet smear.

Exclusion Criteria:

* Women with chlamydia infection, Pregnancy, Herpes

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with vaginal discharge with either bacterial vaginosis or candida infection
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
cure rate | 6 month

SECONDARY OUTCOMES:
colonization of lactobacilli | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Per-Göran Larsson, Principal Investigator — Department of Ob/Gyn Skaraborgs hospital
Locations (2):
- Sweden (2):
  - Department of Ob/Gyn, Skaraborgshospital Skövde, Skövde
  - Kvinnokliniken, Skövde

REFERENCES:
- [Result] Larsson PG, Brandsborg E, Forsum U, Pendharkar S, Andersen KK, Nasic S, Hammarstrom L, Marcotte H. Extended antimicrobial treatment of bacterial vaginosis combined with human lactobacilli to find the best treatment and minimize the risk of relapses. BMC Infect Dis. 2011 Aug 19;11:223. doi: 10.1186/1471-2334-11-223. PMID 21854593
- [Derived] Pendharkar S, Brandsborg E, Hammarstrom L, Marcotte H, Larsson PG. Vaginal colonisation by probiotic lactobacilli and clinical outcome in women conventionally treated for bacterial vaginosis and yeast infection. BMC Infect Dis. 2015 Jul 3;15:255. doi: 10.1186/s12879-015-0971-3. PMID 26137971